CLINICAL TRIAL: NCT01085214
Title: A Phase 2 Study of AZD6244 in Multiple Myeloma
Brief Title: AZD6244 (Selumetinib) in Treating Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02929; NCI-2012-02929 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR669144; NCI-8631; 10-C-0079 (Other: Moffitt Cancer Center); 8631 (Other: CTEP); N01CM00071 (NIH); N01CM00100 (NIH); N01CM62208 (NIH); P30CA076292 (NIH)
Record Dates: First submitted 2010-03-10; First posted 2010-03-11 (Estimated); Results first posted 2015-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-05

CONDITIONS: Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD6244 (Selumetinib) Treatment (Experimental): Participants receive AZD6244 (Selumetinib) orally (PO) twice a day (BID) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Selumetinib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Selumetinib — AZD6244 (Selumetinib), 75 mg was administered orally, twice a day, continuously for 28-day cycles
  Other Names: ARRY-142886; AZD6244; MEK Inhibitor AZD6244

SUMMARY:
This phase II trial studies how well selumetinib works in treating patients with multiple myeloma, a type of cancer in which a specific protein is over active. Selumetinib may stop the growth of cancer cells by blocking this protein.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the response rate of AZD6244 (selumetinib) hydrogen sulfate capsules in patients with relapsed or refractory multiple myeloma (MM).

SECONDARY OBJECTIVES:

I. To evaluate the toxicity of AZD6244 in patients with MM. II. To estimate progression-free survival and duration of response to AZD6244. III. To test whether AZD6244 hydrogen sulfate capsules downregulate tumor cell phosphorylated mitogen-activated protein kinase (pERK)1/2.

OUTLINE:

Patients receive selumetinib orally (PO) twice daily (BID) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of multiple myeloma with relapsed or refractory disease following at least two prior therapies
* Measurable disease defined as:

  * Serum monoclonal protein >= 1 gm/dL or
  * Urine monoclonal protein of >= 200 mg/24 hours, or
  * Measurable free light chains by free light chain assay of >= 10 mg/dL with abnormal kappa to lambda free light chain ratio, or
  * Measurable bone disease, defined as >= 1 unidimensionally measurable lesion (longest diameter to be recorded) >= 20 mm with conventional techniques or >= 10 mm with spiral computed tomography (CT) scan (for patients with lytic bone disease)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Absolute neutrophil count: >= 1,000/μL (independent of blood cell growth factors)
* Platelets: >= 75,000/μL (independent of blood cell growth factors or transfusion)
* Total bilirubin: =< 1.5 x upper normal limit; however, patients with documented Gilbert's syndrome are eligible
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]): < 2.5 x upper limit of normal (ULN)
* Creatinine: < 3.0 x ULN
* Known human immunodeficiency virus (HIV) infected patients meeting the following characteristics are eligible:

  * Cluster of differentiation (CD)4 cell count >= 500/mm^3
  * Meeting either of the following:

    * Willing to suspend antiretroviral therapy for duration of protocol therapy or
    * On stable regimen of combination antiretroviral therapy that does not include either zidovudine or stavudine for at least 12 weeks and without evidence of toxicity
  * No HIV-associated condition that defines acquired immunodeficiency syndrome (AIDS)
* Prior allogeneic stem cell transplant is allowed provided that all of the following conditions are met:

  * >= 6 months have elapsed since allogeneic transplant
  * No graft vs. host disease (GVHD) is present
  * Not currently on immunosuppressive therapy
* Women of child-bearing potential must agree to use a medically accepted form of contraception prior to, during, and for four weeks following study treatment; men must agree to use a medically accepted form of contraception prior to, during, and for sixteen weeks following study treatment
* Able and willing to provide a written informed consent
* Prior palliative and/or localized radiation therapy is permitted, provided at least 14 days have passed from date of last radiation therapy
* Pulse oximetry of >= 95% on room air

Exclusion Criteria:

* Any concurrent condition or planned treatment that would compromise study objectives or represent an unacceptable patient risk, including but not limited to:

  * Planned concurrent treatment for multiple myeloma other than bisphosphonates; ongoing corticosteroids for indications other than multiple myeloma allowed as long as the dose does not exceed 60 mg of prednisone per day or equivalent
  * Persisting effects of any previous or ongoing treatment that might compromise delivery of study treatment or assessment of adverse events
  * Planned concurrent treatment with any other investigational agents
* Cytotoxic chemotherapy less than 2 weeks, or biologic therapy less than 2 weeks, or corticosteroids less than 2 weeks prior to registration
* No other malignancy unless the patient has been disease-free for >= 1 year
* Known multiple myeloma of central nervous system or leptomeninges
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to AZD6244
* Previous mitogen activated protein kinase (MEK) inhibitor use
* Uncontrolled hypertension, i.e., persistent blood pressure (BP) of >= 160/95
* Significant cardiovascular disease (New York Heart Association class II, III or IV cardiac disease), hypertrophic cardiomegaly or restrictive cardiomyopathy, myocardial infarction within the past 6 months, unstable angina, unstable arrhythmia unstable or a need for anti-arrhythmic therapy (use of medication for atrial fibrillation is allowed, if stable for at least 3 months)
* Refractory nausea and vomiting, chronic gastrointestinal diseases (e.g. inflammatory bowel disease), or significant bowel resection that would preclude adequate absorption
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or nursing
* Left ventricular ejection fraction (LVEF) =< 45% by echocardiogram (ECHO) or multigated acquisition scan (MUGA) scan
* Any requirement for supplemental oxygen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Grant, M.D., Principal Investigator — Massey Cancer Center
Locations (9):
- United States (9):
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Mark O Hatfield-Warren Grant Magnuson Clinical Center, Bethesda, Maryland
  - National Institutes of Health, Bethesda, Maryland
  - Billings Clinic Cancer Center, Billings, Montana
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 6 sites in the United States, from April 1, 2010 through July 28, 2011.
Groups:
- AZD6244 (Selumetinib) Treatment: Participants received AZD6244 (Selumetinib) orally (PO) twice a day (BID) on days 1-28. Courses repeated every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | AZD6244 (Selumetinib) Treatment
Started | 37
Completed | 36
Not Completed | 1
Not completed — Alternate treatment required | 1

BASELINE CHARACTERISTICS:
Population: All participants enrolled.
Arm/Group | AZD6244 (Selumetinib) Treatment
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 19
Age, Continuous [Median (Full Range); unit: years] | 65 [43 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall Response: Stringent Complete Response (sCR) + Complete Response (CR) + Very Good Partial Response (VGPR) + Partial Response (PR).
Time Frame: Up to 2 years
Population: All participants who received study treatment
Measure: Number; unit: participants
Arm/Group | AZD6244 (Selumetinib) Treatment
Number analyzed (Participants) | 36
participants
  Response: Total | 2
  Response: sCR | 0
  Response: CR | 0
  Response: VGPR | 1
  Response: PR | 1
  Other Status: Stable Disease | 17
  Other Status: Progressive Disease | 13
  Could not be assessed | 4

2. Secondary Outcome: Duration of Response
Description: Mean duration of response in months. Estimated using the method of Kaplan-Meier.
Time Frame: From response to disease progression or death, assessed up to 2 years
Population: All participants with response
Measure: Mean (Full Range); unit: months
Arm/Group | AZD6244 (Selumetinib) Treatment
Number analyzed (Participants) | 2
months | 4.95 [4.83 to 5.06]

3. Secondary Outcome: Incidence of Toxicity That May Be Treatment Emergent
Description: Participants with Grade 3, 4, and 5 toxicities possibly, probably, or definitely related to study treatment. Toxicity graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE).
Time Frame: 1 year, 11 months
Population: All participants who received study treatment
Measure: Number; unit: participants
Arm/Group | AZD6244 (Selumetinib) Treatment
Number analyzed (Participants) | 36
participants
  Hematologic - Any Grade 3 | 6
  Hematologic - Any Grade 4 | 2
  Hematologic - Any Grade 5 | 0
  Non-Hematologic - Any Grade 3 | 14
  Non-Hematologic - Any Grade 4 | 1
  Non-Hematologic - Any Grade 5 | 3

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Median PFS in months. Progressive Disease (PD): Increase of >= 25% from baseline. Estimated using the method of Kaplan-Meier.
Time Frame: From registration to progression or death, assessed up to 2 years
Population: All participants who received study treatment
Measure: Median (Full Range); unit: months
Arm/Group | AZD6244 (Selumetinib) Treatment
Number analyzed (Participants) | 36
months | 3.52 [2.60 to 5.92]

5. Other Pre Specified Outcome: Changes in Bone Marrow Microenvironment
Description: Effect of AZD6244 on the bone marrow microenvironment in MM.
Time Frame: Baseline to up to 20-30 hours after receiving the first dose of AZD6244
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Level of Key Regulators
Description: The level of key regulators of the MEK/MAPK and PI3K pathways and HSP90 and cell cycle regulators may determine the anti-tumor response to AZD6244 in vivo in multiple myeloma (MM).
Time Frame: Up to 20-30 hours after receiving the first dose of selumetinib
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year, 11 months
Arm/Group | AZD6244 (Selumetinib) Treatment
Serious Adverse Events (participants affected / at risk) | 23/36
Other Adverse Events (participants affected / at risk) | 35/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD6244 (Selumetinib) Treatment (N=36)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Death, NOS (General disorders) | 3 (3)
Flu like symptoms (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Sepsis (Infections and infestations) | 3 (3)
Skin infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3)
CPK increased (Investigations) | 3 (3)
INR increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 5 (7)
Platelet count decreased (Investigations) | 5 (5)
White blood cell decreased (Investigations) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3)
Renal and urinary disorders - Other, Acute renal failure (Renal and urinary disorders) | 1 (1)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Angular cheilitis, unilateral (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD6244 (Selumetinib) Treatment (N=36)
Diarrhea (Gastrointestinal disorders) | 27 (46)
Nausea (Gastrointestinal disorders) | 11 (15)
Vomiting (Gastrointestinal disorders) | 11 (16)
Abdominal pain (Gastrointestinal disorders) | 4 (5)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 18 (29)
Edema, limbs (General disorders) | 16 (20)
Edema, face (General disorders) | 7 (7)
Pain (General disorders) | 4 (4)
Fever (General disorders) | 4 (4)
Localized edema (General disorders) | 4 (6)
Chills (General disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 14 (18)
Neutrophil count decreased (Investigations) | 12 (33)
White blood cell decreased (Investigations) | 12 (29)
Platelet count decreased (Investigations) | 10 (16)
CPK increased (Investigations) | 9 (12)
Alanine aminotransferase increased (Investigations) | 6 (7)
Creatinine increased (Investigations) | 5 (5)
Lymphocyte count decreased (Investigations) | 5 (11)
Alkaline phosphatase increased (Investigations) | 3 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 16 (27)
Hypomagnesemia (Metabolism and nutrition disorders) | 9 (15)
Hypocalcemia (Metabolism and nutrition disorders) | 7 (12)
Hyponatremia (Metabolism and nutrition disorders) | 7 (8)
Hypophosphatemia (Metabolism and nutrition disorders) | 7 (9)
Hypokalemia (Metabolism and nutrition disorders) | 5 (5)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (5)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (4)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (3)
Hypernatremia (Metabolism and nutrition disorders) | 2 (2)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 17 (26)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (6)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 5 (8)
Periorbital edema (Skin and subcutaneous tissue disorders) | 3 (3)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 17 (27)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Sinusitis (Infections and infestations) | 2 (3)
Upper respiratory infection (Infections and infestations) | 2 (2)
Dizziness (Nervous system disorders) | 4 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (8)
Headache (Nervous system disorders) | 2 (3)
Hypertension (Vascular disorders) | 8 (9)
Hypotension (Vascular disorders) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 3 (3)
Renal and urinary disorders - Other (Renal and urinary disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less